CLINICAL TRIAL: NCT05423977
Title: An Open-label, Multicenter, Phase I Dose-escalation Study to Assess the Safety, Pharmacokinetic (PK), Immunogenicity and Preliminary Anti-tumor Activity of ZV0203 in Patients With HER2-Positive Advanced Solid Tumors
Brief Title: Study of ZV0203 in Patients With HER2-Positive Advanced Solid Tumors
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Adcoris Biopharmacy Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZV0203-001CN
Record Dates: First submitted 2022-01-14; First posted 2022-06-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-03

CONDITIONS: HER2-positive Advanced Solid Tumor
Keywords: Advanced Solid Tumor; HER2-positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental:ZV0203 (Experimental)
  Interventions: Drug: ZV0203

INTERVENTIONS:
Drug: ZV0203 — Participants will be allocated to one of the following dose groups: 0.3, 0.6, 1.2, 1.8, 2.7 and 3.6 mg/kg, and receive a treatment of ZV0203-ADC followed by 21 days of dose limited toxicity (DLT) observation period.

SUMMARY:
An open-label, multicenter, phase I dose-escalation study to assess the safety, Pharmacokinetic (PK), immunogenicity and preliminary anti-tumor activity of ZV0203 in patients with HER2-Positive advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Being willing and capable of signing a written informed consent form (ICF).
2. Aged ≥18 or older at the time of signing the ICF.
3. Pathologically diagnosed as having an unresectable locally advanced or metastatic solid tumors, refractory or intolerant to standard therapy, or with no standard therapy available.
4. Having HER2-positive disease, i.e. HER2 positive by in situ hybridization on previously collected tumor tissue and/or immunohistochemistry of 3+.
5. The Eastern Cooperative Oncology Group Performance Status (ECOG) performance status score is 0 or 1.
6. Echocardiography (ECHO) or multi-gated acquisition (MUGA) scan shows a left ventricular ejection fraction of ≥ 50%.
7. Good hematology and end-organ function, with laboratory results within 14 days prior to the first study treatment (Cycle 1, Day 1) meeting the following criteria:

   * Absolute neutrophil count ≥ 1,500/mm3
   * Platelet count ≥ 100,000/mm3 and no transfusion within 14 days after obtaining a hematology laboratory sample at screening
   * Hemoglobin ≥ 9.0 g/dL
   * Total bilirubin ≤ 1.5 ×upper limit of normal (ULN); subjects with confirmed/suspected Gilbert's disease, bilirubin ≤ 3 × ULN
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × ULN; ≤ 5 × ULN if there is liver metastasis
   * Serum creatinine ≤ 1.5 × ULN or estimated glomerular filtration rate > 40 mL/min/1.73 m2
   * Prothrombin time and activated partial thromboplastin time ≤ 1.5 × ULN. It is applicable only to subjects who have received no therapeutic anticoagulant therapy and subjects who have received therapeutic anticoagulant therapy at a stable dose.
8. The investigator determined that the life expectancy of the subjects is ≥12 weeks.
9. For women of childbearing potential, their pregnancy test must be negative for enrollment, and they must agree to take highly effective contraceptive measures when enrolled, during treatment and 90 days after the last dose of the investigational drug (see section 6.1.3). Women are considered to be of childbearing potential from menarche to menopause (after at least 12 months without menstruation) unless they are permanently infertile (due to hysterectomy, bilateral salpingectomy or bilateral oophorectomy).
10. For men, they must be surgically sterile or agree to take highly effective contraceptive measures when enrolled, during treatment and 90 days after the last dose of the investigational drug (see section 6.1.3 ).

Exclusion Criteria:

1. Subjects with symptomatic brain metastases or soft meningeal disease known to require steroid therapy. Subjects diagnosed with brain metastases in the past can participate in the study if they have completed the treatment, recovered from the acute reaction of radiotherapy or surgery prior to enrollment, have discontinued the use of corticosteroids for the treatment of these metastases, and have been clinically stable and neurologically stable without anticonvulsants for at least 4 weeks prior to enrollment.
2. Subjects who are suffering from uncontrolled or major cardiovascular disease, including any of the following circumstances:

   * Baseline QT Interval Corrected Using Fridericia's Formula >450 msec or congenital long QT syndrome.
   * Subjects who have a history of symptomatic congestive heart failure or current symptomatic congestive heart failure (NYHA Grade III-IV) or severe arrhythmias requiring treatment.
   * Subjects who have a history of myocardial infarction or unstable angina within 6 months prior to first dose of ZV0203.
   * Subjects who have a clinically significant resting bradycardia (< 50 beats/min).
   * Subjects who have a history of grade II (Mobitz II) or grade III cardiac conduction block (subjects with pacemakers may participate in this study if they have no history of syncope or clinically relevant arrhythmias during pacemaker use).
   * Subjects who have a history of complete left bundle branch block.
3. Subjects who have a history of clinically significant lung disease (e.g., interstitial pneumonia, pulmonary fibrosis, and severe radiation pneumonia) or suspicion of these diseases by imaging at screening.
4. Subjects who have a history of ocular abnormalities and judged to be ineligible for enrollment by the investigator.
5. Subjects who have received any anticancer treatment or investigational therapy within 4 weeks prior to the first dose of ZV0203.
6. Subjects who have received hormone therapy within 14 days prior to the first dose of ZV0203, except hormone therapy for non-cancer related conditions (e.g. alternative therapies of insulin and hormone for diabetes).
7. Subjects who have undergone major surgery or scheduled surgery for any reason within 4 weeks prior to screening or those the investigator believe may require surgery.
8. Toxicity of prior anticancer therapy does not improve to NCI-CTCAE V5.0 Grade 0 or 1, except for alopecia and laboratory values listed according to the inclusion criteria.
9. Subjects who have a history of other malignancies, except adequately treated non-melanoma skin cancer, radically treated in situ disease or other solid tumors that have been radically treated and free of evidence of disease for at least 2 years.
10. Subjects who are suffering an active infection that is difficult to control with systemic therapy.
11. Subjects who are suffering known active clinically relevant liver disease (e.g., active hepatitis B or active hepatitis C).
12. Subjects who are known to have a history of human immunodeficiency virus infection.
13. Subjects who are suffering a concomitant disease that may increase the risk of toxicity in the judgment of the investigator.
14. Subjects who are known to be allergic to any component of ZV0203.
15. Subjects who have a history of intolerance to pertuzumab or Trastuzumab emtansine (e.g. grade 3 or grade 4 infusion-related reactions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and serious adverse events (SAEs) | From the day of ICF sign to 30 days after the day of the last treatment
  To investigate the safety characteristics.
Maximum Tolerated dose of ZV0203 | 21 days after first treatment
  To determine the maximum tolerated dose (MTD) or the recommended Phase 2 dose (RP2D) of ZV0203.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter of Peak plasma Concentration (Cmax) | 45 days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
Pharmacokinetic (PK) parameter of Peak plasma Concentration (Tmax) | 45 days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
Pharmacokinetic (PK) parameter the area under the plasma concentration-time curve from time zero to the last measurable time point (AUC0-t) | 45 days
  To assess the pharmacokinetic profile in patients with advanced solid tumors
Objective response rate (ORR) | Approximately 1 year
  The objective response rate in patients of advanced solid tumors
Duration control rate (DCR) | Approximately 1 year
  The duration control rate in patients of advanced solid tumors
Duration of response (DOR) | Approximately 1 year
  The duration of response in patients of advanced solid tumors
Progression-free survival (PFS) | Approximately 1 year
  The progression-free survival in patients of advanced solid tumors
Immunogenicity assessment | 45 days
  The endpoints for ZV0203 immunogenicity assessment include the number and percentage of subjects with detectable drug-resistant antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, MD,PhD, Principal Investigator — Peking University Care Luzhong Hospital
Locations (1):
- PKUCare Luzhong Hospital, Zigong, Shandong, China

IPD SHARING:
Plan to Share IPD: No